CLINICAL TRIAL: NCT02185430
Title: Effects of Dexmedetomidine on Respiratory Mechanics and Oxygenation During One Lung Ventilation With Chronic Obstructive Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 4-2014-0306
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: COPD, One Lung Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): saline solution
  Interventions: Drug: saline infusion
- dexmedetomidine group (Active Comparator): dexmedetomidine
  Interventions: Drug: dexmedetomidine infusion

INTERVENTIONS:
Drug: saline infusion — saline infusion, bolus of 1.0 μg kg-1 over 10 min followed by a continuous infusion at 0.5 μg kg-1 h-1 infusion during one-lung ventilation, intravenous
  Arms: Control group
Drug: dexmedetomidine infusion — dexmedetomidine, bolus of 1.0 μg kg-1 over 10 min followed by a continuous infusion at 0.5 μg kg-1 h-1 infusion during one-lung ventilation, intravenous
  Arms: dexmedetomidine group

SUMMARY:
COPD is often associated with the airflow limitation and the pulmonary hyperinflation. During the one-lung ventilation (OLV), COPD patients' physiologic dead space increases and hypercapnia may develop. In addition, an alveolar overdistention by the pulmonary hyperinflation would divert pulmonary blood flow and impair arterial oxygenation. Dexmedetomidine has both vasoconstricting and vasodilatatory effects on a peripheral vasculature and a smooth muscle but its effects on bronchial smooth muscle is unknown. The investigators will evaluate the effects of dexmedetomidine (bolus of 1.0 μg kg-1 over 10 min followed by a continuous infusion at 0.5 μg kg-1 h-1 infusion during one-lung ventilation) as bronchodilator in COPD patients when administered during surgery with the one lung ventilation. If result successfully shows the effect of dexmedetomidine as a predominantly a vasodilator on bronchial tree, the investigators study can support the dexmedetomidine as a vasodilator for pulmonary vessels and bronchial smooth muscle and as an excellent adjunct to anesthetic agents in COPD patients during the OLV.

ELIGIBILITY:
Inclusion Criteria:

1. Above 40 years of age
2. American Society of Anesthesiologists (ASA) Physical Status I, II, III.
3. COPD diagnosed , criteria ( on preop. PFT : FEV1 < 80%, FEV1 / FVC < 70% after bronchodilator)
4. thoracic surgical procedure

Exclusion Criteria:

1. severe functional liver or kidney disease
2. diagnosed HF ( NYHA class >3)
3. arrhythmia or received treatment with antiarrythmic drug .
4. exceed BMI > 30 kg/ m2
5. bradycardia (HR <50 bpm)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The change of the oxygenation | At two-lung ventilation (T1) , 20 min after of one-lung ventilation (T2), 30 mins after Dex or placebo saline infusion (T3), 60 mins after Dex or placebo saline infusion (T4), at the termination of surgery in TLV (T5)
  PaO2/FiO2 ratio

CONTACTS AND LOCATIONS:
Overall Officials: Young Jun Oh, MD,PhD, Principal Investigator — Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine

REFERENCES:
- [Derived] Lee SH, Kim N, Lee CY, Ban MG, Oh YJ. Effects of dexmedetomidine on oxygenation and lung mechanics in patients with moderate chronic obstructive pulmonary disease undergoing lung cancer surgery: A randomised double-blinded trial. Eur J Anaesthesiol. 2016 Apr;33(4):275-82. doi: 10.1097/EJA.0000000000000405. PMID 26716866